CLINICAL TRIAL: NCT02937792
Title: Large Volume Bupivacaine 0.5% Versus Small Volume in Elective Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer in anesthesia department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3 ml bupivacaine
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (No Intervention): one with intrathecal 12.5 mg bupivacaine
- experimental (Experimental): one group with intrathecal 15 mg bupivacaine
  Interventions: Drug: intrathecal 15 mg bupivacaine

INTERVENTIONS:
Drug: intrathecal 15 mg bupivacaine — spinal anesthesia with a large dose of bupivacaine 0.5% in elective caesarean section
  Other Names: large dose spinal
  Arms: experimental

SUMMARY:
To test the safety of high dose spinal in elective CS after prolonged sitting position.

DETAILED DESCRIPTION:
This is a prospective double-blind randomized study, designed to include cases in two groups (using epical program for sample size calculation), one study groups and one control group (parallel). Each group should have at least 30 female patients scheduled for elective caesarean section with a total of 60 cases.

ELIGIBILITY:
Inclusion Criteria:

* Full term pregnant female indicated for the elective section under spinal anesthesia with no history of medical importance

Exclusion Criteria:

* Urgent cases, emergency cases, adverse medical history, anticoagulant treatment, associated pregnancy complication, failed spinal, surgical complication or refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
vital signs | 45 minutes
  blood pressure, heart rate

SECONDARY OUTCOMES:
complications | 45 minutes
  nausea, vomiting and total spinal

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided